CLINICAL TRIAL: NCT04101136
Title: Effect of Atorvastatin on Subclinical Atherosclerosis in Virally-suppressed HIV-infected Patients With CMV Seropositivity: a Randomized Double-blind Placebo-controlled Trial
Brief Title: Effect of Atorvastatin on Subclinical Atherosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Evy Yunihastuti, Allergy- Immunology Consultant, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-03-0272; KET-265/UN2.F1/ETIK (Registry Identifier: Ethical Approval)
Record Dates: First submitted 2019-08-28; First posted 2019-09-24 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: CMV
Keywords: statin; atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Atorvastatin tablets in generic form. The placebo tablets will be prepared by Cipto Mangunkusumo hospital pharmacist, were composed of starch and were similar to atorvastatin tablets in size, shape, and colour. The participants will get the medication supply every month along with the refill of antiretroviral drugs. The drug and placebo tablets will be administered to patients by a staff member who are privy to the treatment. In the end of every month, each participant should return the unused pills every month.
Who Masked: Participant, Care Provider
Masking Description: Subjects with undetectable HIV-RNA, positive anti-CMV, having Framingham Risk Score above 10% with LDL < 130 or under 10% with LDL <160 will undergo thorough medical history and anthropometric examination as the initial data. Patient will be seen for regular clinical follow up as standard of care in the clinic (monthly/ bimonthly). Follow up visit will include clinical and laboratory procedure. At week 24, blood collection procedures and neurocognitive examination procedures will be repeated. At week 48, blood collection procedures, CIMT, FMD, transient elastography with CAP, and neurocognitive examination procedures will be repeated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin 20 mg (Active Comparator): Study pharmacist will make code (A and B) for atorvastatin and placebo, then save the code in safe place. Pharmacist will record each subject as participant received A or B intervention.
  Interventions: Drug: Atorvastatin - placebo controlled clinical trial
- Placebo 20 mg (Placebo Comparator): The placebo tablets will be prepared by Cipto Mangunkusumo hospital pharmacist, were composed of starch and were similar to atorvastatin tablets in size, shape, and colour.
  Interventions: Drug: Atorvastatin - placebo controlled clinical trial

INTERVENTIONS:
Drug: Atorvastatin - placebo controlled clinical trial — The participants will get the medication supply every month along with the refill of antiretroviral drugs. The drug and placebo tablets will be administered to patients by a staff member who are privy to the treatment. In the end of every month, each participant should return the unused pills every month
  Other Names: Ator-Placebo

SUMMARY:
Statin administration is supposed to reduce subclinical atherosclerosis by decreasing LDL cholesterol levels, possibly via lipid-independent anti-inflammatory effect. Its pleiotropic properties also adding beneficial effect against CMV infection.

The investigators plan to study atorvastatin in virally- suppressed HIV-infected patients on stable ART with CMV seropositive and statin-naïve to evaluate the subclinical atherosclerosis changes assessed by carotid intima media thickness (CIMT).

DETAILED DESCRIPTION:
Extended description of the protocol, including more technical information

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20 to 45 years old
* Using stable ART at least 1 year
* Positive IgG CMV
* Viral load HIV RNA <50 copies / ml

Exclusion Criteria:

* Undergoing hepatitis C DAA therapy
* Decompensated cirrhosis or acute liver failure
* History of coronary artery disease
* Diabetes mellitus
* History of of brain infection, epilepsy, stroke
* History of rhabdomyolysis or myopathy
* Pregnant or breastfeeding
* Severe depression
* Using statin therapy in the past 6 weeks
* History of statin hypersensitivity
* Framingham Risk Score above 10% within LDL ≥130
* Framingham Risk Score under 10% within LDL ≥160
* Out of Periodontitis Index (Upper right molars, top series, upper left molars, lower right molars, bottom series, lower left molars)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Carotid intima medial tunica change | (1) 0-week visit, (2) 48-week visit
  Numerical changes (in millimeter) between baseline and 48 weeks. Common Carotid Artery (CCA) intima media thickness measured by using B mode imaging system (Affiniti 70 series), equipped with a linear array transducer > 7 MHz with minimal compression (<10:1) and footprint of at least 3 cm. This procedure is operated by certified Cardiologist.
  Reference Siomva I. Intima-media thickness: appropriate evaluation and proper measurement, described. ESC. May 2015;15:21.

SECONDARY OUTCOMES:
Flow mediated vasodilatation change | (1) 0-week visit, (2) 48-week visit
  Numerical changes (in percentage) between baseline and 48 weeks FMD.
  Using a high-resolution ultrasound linear array transducer, longitudinal images of the right brachial artery (mostly 3-15 cm above the elbow) were recorded at the baseline and for 3 minutes after cuff deflation following suprasystolic compression (50 mmHg over the systolic blood pressure) of the right forearm for 5 minutes. This procedure is operated by certified cardiologist.
  Reference:
  Charakida M, Masi S, Luscher TF, Kastelein JJ, Deanfield JE.Assessment of atherosclerosis: the role of flow-mediated dilatation.Eur Heart J. 2010 Dec;31(23):2854-61
Liver fibrosis change | (1) 0-week visit, (2) 48-week visit
  Numerical changes (in KPa) between baseline and 48 week. The measurement of liver stiffness which uses the velocity of shear waves that travel through the liver using the Fibroscan (Echosens) device. This procedure is operated by certified hepatologist.
Liver steatosis change | (1) 0-week visit, (2) 48-week visit
  Numerical changes (in dB/m) between baseline and 48 weeks. The measurement of steatosis using the Fibroscan (Echosens) equipped with CAP software. dB/m. This procedure is operated by certified hepatologist.
Fasting lipid change | (1) 0-week visit, (2) 48-week visit
  Numerical changes of fasting lipid profile consist of total cholesterol, LDL-C, HDL-C and triglyceride in mg/dL. Range of fasting is 8 - 10 hours. The test is located in Cipto Mangunkusumo Hospital or Prodia Laboratory Clinic.
Neurocognitive function change | (1) 0-week visit, (2) 24-week visit, (3) 48-week visit
  Mean or median changes of neurocognitive function change. Neurologist will do supervision while subject do the test. The measurement tool is questionnaire named "neurocognitive test". This item will comprising several aspects:
  1. Trail making test
  2. Symbol digit modalities test
  3. Brief visuospatial memory test revised
  4. California verbal learning test II
Community Periodontal Index (CPI) | (1) 0-week visit, (2) 48-week visit
  This Community Periodontal Index takes into consideration 10 teeth in the oral cavity i.e. 17, 16, 11, 26, 27, 37, 36, 31, 46 and 47 and subsequently evaluates the occurrence of gingival bleeding, presence of supra- and subgingival calculus, periodontal pockets with probing depths between 3.5-6.0 mm, as well as clinical attachment loss. This procedure done by dentist.
  CPI score:
  * Score 0: health periodontal conditions
  * Score 1: gingival bleeding on probing
  * Score 2: calculus and bleeding
  * Score 3: periodontal pocket 4-5 mm
  * Score 4: periodontal pocket ≥6 mm Only the worst ﬁnding from the index teeth is recorded per sextant of teeth.
beta 2-microglobulin change | (1) 0-week visit, (2) 48-week visit
  The numerical change of beta 2-microglobulin (in pg/mL) between 0-week visit and 48-week visit. This examination located in Indonesian Medical Education and Research Institute (IMERI) laboratory
Soluble CD14 change | (1) 0-week visit, (2) 48-week visit
  The numerical change of sCD14 (in pg/mL) between 0-week visit and 48-week visit. This examination located in Indonesian Medical Education and Research Institute (IMERI) laboratory
ICAM-1 change | (1) 0-week visit, (2) 48-week visit
  The numerical change of ICAM-1 (in pg/mL) between 0-week visit and 48-week visit. This examination located in Indonesian Medical Education and Research Institute (IMERI) laboratory
High Sensitivity C-Reactive Protein (hsCRP) change | (1) 0-week visit, (2) 48-week visit
  The numerical change of hsCRP (in mg/L) between 0-week visit and 48-week visit. This examination located in Indonesian Medical Education and Research Institute (IMERI) laboratory
Vascular Cell Adhesion Molecule-1 (V CAM-1) change | (1) 0-week visit, (2) 48-week visit
  The numerical change of V CAM-1 (in pg/mL) between 0-week visit and 48-week visit. This examination located in Indonesian Medical Education and Research Institute (IMERI) laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta, Center Jakarta, Indonesia

REFERENCES:
- [Result] Chastain DB, Stover KR, Riche DM. Evidence-based review of statin use in patients with HIV on antiretroviral therapy. J Clin Transl Endocrinol. 2017 Feb 22;8:6-14. doi: 10.1016/j.jcte.2017.01.004. eCollection 2017 Jun. PMID 29067253
- [Derived] Yunihastuti E, Rusdi L, Syahrir Azizi M, Estiasari R, Jasirwan COM, Wulandari EAT, Purnamasari D, Shinta Noviar M, Aman Nasution S. Effect of atorvastatin on subclinical atherosclerosis in virally-suppressed HIV-infected patients with CMV seropositivity: a randomized double-blind placebo-controlled trial. F1000Res. 2023 Sep 15;10:151. doi: 10.12688/f1000research.28262.2. eCollection 2021. PMID 37772075
- See also: Chastain DB, Kayl RS, Daniel MR. Evidence-based review of statin use in patients with HIV on antiretroviral therapy. J Clin Transl Endocrinol. 2017;8:6-14. — https://www.ncbi.nlm.nih.gov/pubmed/29067253

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04101136/Prot_SAP_000.pdf